CLINICAL TRIAL: NCT05798897
Title: A Phase 1 Study of Patient-Derived Multi-Tumor-Associated Antigen-Specific T Cells (MT-601) Administered to Patients With Relapsed or Refractory Non-Hodgkin and Hodgkin Lymphoma (APOLLO)
Brief Title: Safety and Preliminary Efficacy of MT-601 in Patients With Relapsed/Refractory Lymphoma
Acronym: APOLLO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Marker Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRKR-22-601-01
Record Dates: First submitted 2023-03-14; First posted 2023-04-05 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Non-Hodgkin Lymphoma, Adult; Non-Hodgkin Lymphoma, Refractory; Non-Hodgkin Lymphoma, Relapsed; Non Hodgkin Lymphoma; Hodgkin Lymphoma; Hodgkin Lymphoma, Adult; Hodgkin's Lymphoma, Relapsed, Adult
Keywords: NHL; Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Hodgkin Disease; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): Single arm study evaluating MT-601 investigational product at 200 million cells and 400 million cells per dose
  Interventions: Drug: MT-601

INTERVENTIONS:
Drug: MT-601 — Multi-antigen specific CD4+ andCD8+ T cells

SUMMARY:
This study is a Phase 1 multicenter study with a Dose Escalation and Dose Expansion evaluating safety and efficacy of MT-601 administration to patients with Relapsed or Refractory Lymphoma. The starting dose administered is 200 x 10^6 cells (flat dosing).

DETAILED DESCRIPTION:
This study is a Phase 1, multicenter, open-label study designed to evaluate the safety and efficacy of MT-601 in participants with relapsed or refractory (R/R) non-Hodgkin lymphoma (NHL) or Hodgkin lymphoma (HL) who either relapsed or had incomplete response after cluster of differentiation (CD) 19-directed chimeric antigen receptor (CAR) T cell therapy or are CAR T cell therapy naïve (ineligible or refused CD19-directed CAR T cell therapy or for whom CAR T cell therapy is not available). The study will consist of two portions or phases: 1) Dose Escalation with allowance for backfilling cohorts (up to 50 participants) followed by 2) Dose Expansion at the preliminary RP2DS in 1-2 disease specific cohorts of up to 29 participants each. The Dose Expansion portion of this study will begin after completion of the Dose Escalation portion. The purpose of the Dose Expansion portion of the study is to evaluate the clinical efficacy of MT-601 at the dose determined to be safe in the Dose Escalation portion.

ELIGIBILITY:
Inclusion Criteria:

* All applicable inclusion and exclusion criteria must be met at Screening and at Baseline (re-assessment of eligibility within 14 days prior to group assignment).

Participants are eligible to be included in the study only if all of the following criteria apply and the participant, in the judgement of the Investigator, is an appropriate candidate for experimental therapy:

General:

1. Participant must be ≥ 18 years of age and capable of giving signed informed consent (ICF), which includes compliance with the requirements and restrictions listed in the ICF and in the protocol, at the time of signing the ICF.

   Disease Specific:
2. Cytologically or histologically confirmed diagnosis of NHL, HL or CLL based on the 2022 World Health Organization (WHO) criteria for hematolymphoid neoplasms
3. Enrollment of the following subtypes will be eligible:

   1. LBCL including diffuse large B cell lymphoma, primary mediastinal B cell lymphoma (PMBCL), high grade B cell lymphoma (HGBL), T cell rich B cell lymphoma and transformed indolent lymphoma (transformed iNHL)
   2. FL
   3. MCL
   4. MZL
   5. HL

      The following additional subtypes may be enrolled in disease specific cohorts during Dose Expansion (upon approval by Sponsor)
   6. CLL/SLL
   7. CNS lymphoma
   8. CAR T cell refractory
4. Must have measurable disease as per 2014 Lugano criteria or 2018 iwCLL criteria. Participants with splenic MZL must have measurable splenomegaly on imaging or evidence of bone marrow involvement.

   Prior Treatments
5. Participants who are R/R, are intolerant to, or are considered ineligible for systemic standard of care anticancer treatments, including at least 2 prior therapies. Participants who refuse standard of care treatments may also be considered if documentation is provided that he/she has been made aware of all therapeutic options.
6. For participants with LBCL, FL, and MCL: Have received CD19-directed CAR T cell therapy and relapsed ≥ 30 days or attained an incomplete response as the best response within 1 year after CAR T cell administration. Participants who refuse or are ineligible for CAR T cell therapy are eligible for this study. Note: during Dose Expansion, a specific cohort may be enrolled to evaluate participants who were refractory to CD19-directed CAR T cell therapy.

   Health Status
7. Karnofsky score of ≥70 or performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
8. Life expectancy ≥12 weeks
9. Adequate blood, liver, renal and cardiac function:

   1. Hematology: Hemoglobin ≥ 7.0 g/dL (can be transfused), absolute lymphocyte count (ALC) ≥ 300/μL, (prior to apheresis only), absolute neutrophil count (ANC) ≥ 750/μL and platelet count ≥ 50,000/μL (prior to the conditioning regimen only)
   2. Liver: Bilirubin ≤ 1.5X upper limit of normal (ULN) (exception of bilirubin elevation due to Gilbert's syndrome 3X); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3X ULN
   3. Renal: Serum creatinine ≤ 1.5X ULN or measured or calculated creatinine clearance ≥ 50 mL/min (prior to the conditioning regimen)
   4. Cardiac: left ventricular ejection fraction ≥ 45% (prior to the leukapheresis) Sex
10. Female: Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective (i.e., with a failure rate of < 1% per year), preferably with low user dependency during the intervention period and for at least 6 months after the last infusion of MT-601 and agrees not to donate eggs (i.e., ova and oocytes) for the purpose of reproduction during this period
11. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 6 months after the last infusion of MT-601:

Refrain from donating sperm

PLUS either:

Be abstinent from intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR Must agree to use a male condom AND should also be advised of the benefit for a nonpregnant female partner to use a highly effective method of contraception as a condom may break or leak

Exclusion Criteria:

* Patients are excluded from the study if any of the following criteria apply:

Disease-related

1. Evidence of bulky disease at the time of the conditioning regimen (≥ 10 cm in diameter for LBCL or HL and > 6 cm for other subtypes)
2. Untreated or ongoing treatment for CNS lymphoma or completed treatment within 2 weeks of apheresis (Note: May be allowed in Dose Expansion if disease specific cohort for CNS lymphoma is opened)
3. Refractory to CAR T therapy defined as a best response of stable disease or disease progression (Note: May be allowed in Dose Expansion if disease specific cohort for CAR T cell therapy refractory is opened)
4. Requirement for urgent therapy due to tumor mass effects such as bowel obstruction or blood vessel compression Medical Conditions
5. Primary immunodeficiency
6. Severe or uncontrolled autoimmune disorder
7. History or presence of clinically relevant CNS pathology such as epilepsy, seizure, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
8. Unresolved immune effector cell-associated neurotoxicity syndrome (ICANS) from prior CAR T cell administration. Consideration for Grade 1 may be made after discussion with the Medical Monitor
9. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g., cervix, bladder, breast, and/or prostate) unless disease free for at least 3 years
10. Cardiac conditions:

    1. Medically uncontrolled hypertension (≥ 160 mmHg systolic blood pressure or ≥ 100 mmHg diastolic blood pressure)
    2. Congestive heart failure Class ≥ II as defined by the New York Heart Association
    3. Acute coronary syndrome (including unstable angina, coronary artery stenting, or angioplasty, bypass grafting within prior 6 months)
    4. History or evidence of current, uncontrolled, clinically significant, unstable arrhythmias
11. Oxygen saturation at room air < 92%
12. Participant has known human immunodeficiency virus (HIV) infection, or active hepatitis B virus (HBV)/hepatitis C virus (HCV) infection
13. Acute bacterial, viral, fungal infection requiring systemic therapy (uncomplicated urinary tract infection and bacterial pharyngitis are permitted if responding to therapy)
14. History of severe allergic reactions to any of the study intervention components including conditioning regimen, dimethyl sulfoxide (DMSO) or to tocilizumab
15. Clinically significant reversible toxicities from prior cancer therapy that have not recovered to Grade 1 or baseline

    * Participants with Grade 2 neuropathies due to prior treatment will be allowed on study.
    * Participants with clinical nonsignificant toxicities, such as alopecia, will be allowed on study.

    Prior/Concomitant Therapy

    Prior to Apheresis:
16. Receipt of allogeneic hematopoietic cell transplant (HCT) within 12 months; on immunosuppression or with evidence of donor/mixed chimera
17. Receipt of autologous HCT within 3 months
18. Treatment with CD19-directed CAR T cell therapy within 3 months
19. Treatment with bispecific antibody within 1 month
20. Treatment with antibody drug conjugates (ADC's) or PD-1/PD-L1 within 21 days
21. Treatment with monoclonal antibodies impacting T cell function within 14 days
22. Treatment with systemic immunosuppression including systemic corticosteroids (unless ≤5 mg/day oral prednisone or steroid equivalent) within 14 days
23. Treatment with chemotherapy within 7 days

    Prior to the conditioning regimen:
24. Treatment with a live, attenuated vaccine within 4 weeks
25. Treatment with antibody drug conjugates (ADC's) or PD-1/PD-L1 within 21 days
26. Treatment with chemotherapy or biologics/monoclonal antibodies within 14 days
27. Treatment with radiation therapy within 7 days
28. Treatment with a tyrosine kinase inhibitor (TKI) within 7 days or 5 half-lives (whichever is longer) before conditioning regimen
29. Hematopoietic growth factors <2 days

    At either time:
30. Treatment with experimental CAR T cell product unless approved by Medical Monitor
31. Treatment with other cancer therapy including investigational agents that do not fit in the above categories within 14 days
32. Major surgery within 14 days

    Other
33. Pregnant or lactating
34. Any other issue which, in the opinion of the treating physician, would make the participant ineligible for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation | After 3 or 6 patients in each dose cohort have been treated with MT-601 and have had the opportunity to be followed for 28 days.
  To assess safety and tolerability of escalating doses of MT-601 by the number of participants with MT-601 Dose Limiting Toxicities (DLTs) and Safety events (including but not limited to): treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), deaths, and clinical laboratory abnormalities per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Dose Expansion (ORR) | 12 months after the last patient treated in the Dose Expansion portion of the study receiving the first dose of MT-601.
  To assess anti-tumor activity of MT-601 based on Lugano Classification by the following endpoints:
  * Objective response rate (ORR) defined as the proportion of treated patients who achieve a best response of complete remission (CR) or partial response (PR) per Lugano Classification.
  * The Clopper-Pearson method will be used to estimate the two-sided exact 95% confidence interval for ORR.
Dose Expansion (DOR) | 12 months after the last patient treated in the Dose Expansion portion of the study receiving the first dose of MT-601.
  To assess anti-tumor activity of MT-601 based on Lugano Classification by the following endpoints:
  * Duration of response (DOR) defined for patients who attain a best response of CR or PR and is the time between the date of first documented CR or PR and the date of the first observed progression per Lugano Classification.
  * DOR will be estimated using the Kaplan-Meier (KM) product limit method. The median DOR and corresponding 95% confidence intervals (CI) will be estimated.
Dose Expansion (CR) | 12 months after the last patient treated in the Dose Expansion portion of the study receiving the first dose of MT-601.
  To assess anti-tumor activity of MT-601 based on Lugano Classification by the following endpoints:
  * Complete remission (CR) rate defined as the proportion of treated patients who achieve a best response of CR per Lugano Classification.
  * The Clopper-Pearson method will be used to estimate the two-sided exact 95% confidence interval for CR rate estimates.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - University of Colorado, Aurora, Colorado
  - Colorado Blood Cancer Institute (Sarah Cannon), Denver, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cornell, New York, New York
  - Sarah Cannon Research Institute at St. David's South Austin, Austin, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No